CLINICAL TRIAL: NCT06942260
Title: Vascular Access Registry (VARegistry) - Prospective Registry of Vascular Access
Brief Title: Vascular Access Registry
Acronym: VARegistry
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Grigorios Tsigkas, Associate Professor of Cardiology, University Hospital of Patras
Other Study IDs: 362/05.09.2024
Record Dates: First submitted 2025-03-11; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Vascular Access; Coronary Interventions
Keywords: Vascular Access; Coronary Interventions; Coronary Angiography; Radial Artery; Distal Radial Artery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Radial Artery Approach
- Distal Radial Artery Approach
- Femoral Artery Approach
- Ultrasound-Guided Radial Artery Approach
- Ultrasound-Guided Distal Radial Artery Approach
- Ultrasound-Guided Femoral Artery Approach

SUMMARY:
The Vascular Access Registry (VARegistry) is a prospective patient registry that will be conducted at the Hemodynamic Laboratory of the Cardiology Clinic of the University General Hospital of Patras.

The puncture of the vessel will be performed either using palpation, anatomical landmarks or using ultrasound guidance, depending on the ability and preference of each operator. Patients who meet all admission criteria and no exclusion criteria will be admitted to the study.

Patients >18 years of age presented with indication for any percutaneous cardiac procedure will be included in the study. No exclusion criteria exist.

The vascular puncture will be performed according to current guidelines and on the basis of recent scientific data. If the attempt to obtain access from the selected location is unsuccessful, the access location will be changed. The choice of the new access location in case of failure of the originally selected one is subject to the preference of each operator.

Participants will be monitored for the period they remain hospitalized, depending on the initial indication of intervention, and a follow-up with a vascular ultrasound after one month is recommended.

The primary endpoint is the percentage of success of the puncture at the initial access point.

The secondary endpoints are as follows:

* Percentages of successful puncture of vascular access with and without the use of ultrasound guidance
* Occlusion rate of the access artery before discharge
* Crossover rate of access site during procedure
* Time to sheath placement during procedure
* Total intervention time
* Procedure duration (from the sheath insertion to the completeness of the procedure)
* Total fluoroscopy time
* Total DAP (Dose area product)
* Air Kerma
* Time required for hemostasis
* Vascular complications *
* Classification of hematomas (modified classification by EASY)**
* Vascular implication of access artery using ultrasound monitoring of patients at 30 days

  * VARC criteria ** if the forearm has been used

DETAILED DESCRIPTION:
A. Introduction Ensuring vascular access is a prerequisite for coronary angiography and/or angioplasty (Percutaneous Coronary Intervention - PCI), and for transcatheter aortic valve replacement (TAVR). Femoral access has been the established access route for several decades regarding coronary interventions and currently for structural heart disease, mainly due to the size of the sheaths. However, due to increased vascular complications, speaking mostly for coronary interventions, alternative access routes with additional benefits have been sought. In this context, the brachial artery and the ulnar artery were tested without the expected results, while the radial artery presented the most favourable characteristics and was eventually established as the main access route. Recent guidelines from the European Heart Society (ESC), the American College of Cardiology (ACC), American Heart Association (AHA) and the Society for Cardiovascular Angiography and Interventions (SCAI) recommend the TransRadial Approach (TRA) for both acute and chronic coronary syndromes, as well as complex coronary interventions.

Recently, an alternative transradial approach through the anatomical snuffbox has been proposed. Large, randomized studies have shown that the distal TransRadial Approach (dTRA) is a safe method, with faster hemostasis time and lower rates of obstruction of the radial artery. (Radial Artery Occlusion - RAO). Initially, it was shown that dTRA reduces the rate of RAO in the forearm, compared to TRA in the first 1-30 days after intervention. Then, the lower rate of RAO in the dTRA group was confirmed, and the significantly less time required for haemostasis in the dTRA access group was highlighted. The most recent, multicenter study, DISCO-RADIAL, did not show a statistically significant advantage in avoiding RAO when using dTRA, however, it should be noted that RAO prevalence was less than 1% in both access sites.

Both studies showed a lower risk of EASY ≥II hematoma, but ANGIE study showed a statistically significant difference in the incidence of hematomas at the puncture site using a modified EASY scale. There was consensus both on the frequency of crossover of access site from dTRA, and on the longer duration required for gaining access of the dTRA.

A common point of the randomized studies that have been conducted so far is the exclusion of patients with ST-elevation myocardial infarction (STEMI), as the safety and effectiveness of the technique had to be firstly demonstrated, and when the necessary experience was acquired in more stable clinical contexts, it could then be tested in more urgent situations. Similarly, in the case of TRA, STEMI patients were the last framework in which its superiority over the femoral access was proven. Limited data exists to date on the use of dTRA in patients with STEMI, and those are derived from retrospective and prospective studies. In addition, non-randomized studies have shown that dTRA is a reliable alternative to TRA and femoral approach in the emergency setting. Nevertheless, no randomized studies have yet been published comparing dTRA with TRA in STEMI patients.

Despite the increasing use of transradial access and consequential reciprocal reduction in femoral access use for coronary angiography and PCI, femoral access remains necessary for numerous procedures, many of which require large-bore access. The transfemoral approach is the preferred and most commonly used access for transcatheter aortic valve replacement. Femoral access is used in most cases of mechanical circulatory support, such as in the setting of cardiogenic shock, cardiac arrest, or high-risk PCI with such devices as intra-aortic balloon pump, Impella (Abiomed, Danvers, Massachusetts), or venoarterial extracorporeal membrane oxygenation. Additionally, femoral access is preferred for some complex coronary interventions, such as coronary chronic total occlusion PCI.

Finally, although ultrasound guidance for vascular access has been widely adopted, its use for gaining transradial access in the cardiac catheterization laboratory is rare, even though data show an improvement in the success rates of obtaining radial access.

B. Objective The purpose of VARegistry is to evaluate the safety and effectiveness of any vascular access used in daily clinical practice for percutaneous cardiac interventions, with emphasis on access from the distal radial artery (DRA) both anatomically and using ultrasound.

VARegistry seeks to answer critical questions about the success rates of cardiac procedures through vascular access and to record any complications from the various vascular access points. Moreover, the frequency of vascular obstruction is recorded, the frequency of bleeding and other local or systemic interventional complications, in an attempt to define the factors affecting the success of the puncture.

C. Study Design The Vascular Access Registry (VARegistry) is a prospective patient registry that will be conducted at the Hemodynamic Laboratory of the Cardiology Clinic of the University General Hospital of Patras.

The puncture of the vessel will be performed either using palpation, anatomical landmarks or using ultrasound guidance, depending on the ability and preference of each operator. Patients who meet all admission criteria and no exclusion criteria will be admitted to the study.

The protocol of the study will be approved by both the Scientific and Ethics Committees of the conducting hospital, and will also be registered at clinicaltrial.gov.

C.1 Study population and monitoring Patients >18 years of age presented with indication for any percutaneous cardiac procedure will be included in the study (Table 1). The exclusion criteria are presented in Table 1.

Participants will be monitored for the period they remain hospitalized, depending on the initial indication of intervention, and a follow-up with a vascular ultrasound after one month is recommended.

Admission Criteria Age>18 years Indication for percutaneous cardiac procedure

Exclusion Criteria No exclusion criteria exist Table 1. Admission and exclusion criteria

Patients who meet the admission criteria will participate in the study. The researchers will inform the patients about the purpose of the study, the procedures to be followed and the estimated duration. Each patient will be informed that their participation is voluntary and can withdraw from the study at any time, without any impact on their treatment. The patient will be informed that his/her medical data may be examined by authorized staff. All patients need to provide signed approval to participate in the study. The initial consent of the patient before the catheterization, can be oral. If the patient orally agrees to participate in the study, written consent will follow. A copy of the written consent will then be given to the patient and the original will be kept in the study records.

C.2 Vascular access procedure The vascular puncture will be performed according to current guidelines and on the basis of recent scientific data. If the attempt to obtain access from the selected location is unsuccessful, the access location will be changed. The choice of the new access location in case of failure of the originally selected one is subject to the preference of each operator.

C.3 Hemostasis protocol After the intervention is completed, any hemostasis device available in the hemodynamic laboratory can be used. The access site is examined for hemostasis in 30 minutes, 1, 2 and 3 hours from the moment the device was set, and if not achieved within this timeframe, manual compression is applied.

C.4 Sample population Based on a pilot recording program, which started in December 2023 and to which ultrasound guidance was introduced in May 2023, where 1,157 patients were admitted to the study (over a period of 18 months), the investigators estimate a similar sample-size of patients in a 18-month prospective registry that will begin on 1/1/2025 and end on 30/6/2026.

D. End Points The primary endpoint is the percentage of success of the puncture at the initial access point during the procedure.

The secondary endpoints are as follows:

* Percentages of successful puncture of vascular access with and without the use of ultrasound guidance
* Occlusion rates of the access artery before discharge
* Crossover rate of access site during procedure
* Time to sheath placement
* Total intervention time
* Procedure duration (from the sheath insertion to the completeness of the procedure)
* Total fluoroscopy time
* Total DAP (Dose area product)
* Air Kerma
* Time required for hemostasis
* Type and rate of vascular complications until hospital discharge *
* Classification of hematomas (modified classification by EASY)**
* Type and rate of vascular implications of access artery using ultrasound monitoring of patients at 30-day follow-up

  * VARC criteria (Figure 1) ** if the forearm has been used

E. Quality control and personal data protection The training of the principal investigator and other research staff who will participate in the study is the responsibility of the study's principal investigator.

All research staff involved in the study will be guided by the invasive cardiologist who has been selected as the principal investigator at the respective centre. Independent supervision will be carried out throughout the study in accordance with Good Clinical Practice (GCP).

The data is imported by the researcher in a special eCRF. There are standard operating procedures and regular full backups to ensure that data will not be lost and that it can be recovered in case of equipment failure, (unintentional) data destruction or destruction.

F. Conclusion The present prospective study aims to highlight the tendency of modern invasive cardiologists to constantly approach smaller arteries, where this is feasible. In addition, it seeks to explore the potential benefits that the use of ultrasound-guided puncture can have in daily clinical practice, regardless of the vascular access point.

ELIGIBILITY:
Inclusion Criteria:

* Indication for percutaneous cardiac procedure

Exclusion Criteria:

* No exclusion criteria exist

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients >18 years of age presented with indication for any percutaneous cardiac procedure will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1157 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of success of the puncture at the initial access point | From puncture of access site until successful sheath insertion

SECONDARY OUTCOMES:
Percentages of successful puncture of vascular access with and without the use of ultrasound guidance | Until successful sheath insertion
Occlusion rate of the access artery before discharge | From the completion of procedure until hospital discharge
Crossover rate of access site during the procedure | From first puncture of primary access site until successful sheath insertion
Time to sheath placement | From first puncture of primary access site until successful sheath insertion
Total intervention time | From first puncture of primary access site until successful completion of the procedure
Procedure duration | From the sheath insertion to the completeness of the procedure
Total fluoroscopy time | From the sheath insertion to the completion of the procedure
Total DAP (Dose area product) | From the sheath insertion to the completion of the procedure
Air Kerma | From the sheath insertion to the completion of the procedure
Time required for hemostasis | From the application of any hemostasis device until hemostasis is achieved
Type and rate of vascular complications before discharge | From the start of the procedure until hospital discharge
Classification of hematomas | From the start of the procedure until hospital discharge
Type and rate of vascular implications of access artery using ultrasound monitoring until follow-up | From the start of the procedure until 30-day follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department, University Hospital of Patras, Pátrai, ACHAIA, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mason PJ, Shah B, Tamis-Holland JE, Bittl JA, Cohen MG, Safirstein J, Drachman DE, Valle JA, Rhodes D, Gilchrist IC; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Peripheral Vascular Disease; and Council on Genomic and Precision Medicine. An Update on Radial Artery Access and Best Practices for Transradial Coronary Angiography and Intervention in Acute Coronary Syndrome: A Scientific Statement From the American Heart Association. Circ Cardiovasc Interv. 2018 Sep;11(9):e000035. doi: 10.1161/HCV.0000000000000035. PMID 30354598
- [Background] Tsigkas G, Moulias A, Papageorgiou A, Ntouvas I, Grapsas N, Despotopoulos S, Apostolos A, Papanikolaou A, Smaili K, Vasilagkos G, Davlouros P, Hahalis G. Transradial access through the anatomical snuffbox: Results of a feasibility study. Hellenic J Cardiol. 2021 May-Jun;62(3):201-205. doi: 10.1016/j.hjc.2020.02.002. Epub 2020 Mar 2. PMID 32135274
- [Background] Didagelos M, McEntegart M, Kouparanis A, Tsigkas G, Koutouzis M, Tsiafoutis I, Kassimis G, Oldroyd KG, Ziakas A. Distal Transradial (Snuffbox) Access for Coronary Catheterization: A Systematic Review. Cardiol Rev. 2021 Jul-Aug 01;29(4):210-216. doi: 10.1097/CRD.0000000000000339. PMID 34061817
- [Background] Sgueglia GA, Hassan A, Harb S, Ford TJ, Koliastasis L, Milkas A, Zappi DM, Navarro Lecaro A, Ionescu E, Rankin S, Said CF, Kuiper B, Kiemeneij F. International Hand Function Study Following Distal Radial Access: The RATATOUILLE Study. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1205-1215. doi: 10.1016/j.jcin.2022.04.023. Epub 2022 May 17. PMID 35595672
- [Background] Sgueglia GA, Lee BK, Cho BR, Babunashvili A, Lee JB, Lee JW, Schenke K, Lee SY, Harb S. Distal Radial Access: Consensus Report of the First Korea-Europe Transradial Intervention Meeting. JACC Cardiovasc Interv. 2021 Apr 26;14(8):892-906. doi: 10.1016/j.jcin.2021.02.033. PMID 33888235
- [Background] Eid-Lidt G, Rivera Rodriguez A, Jimenez Castellanos J, Farjat Pasos JI, Estrada Lopez KE, Gaspar J. Distal Radial Artery Approach to Prevent Radial Artery Occlusion Trial. JACC Cardiovasc Interv. 2021 Feb 22;14(4):378-385. doi: 10.1016/j.jcin.2020.10.013. PMID 33602433
- [Background] Tsigkas G, Papageorgiou A, Moulias A, Kalogeropoulos AP, Papageorgopoulou C, Apostolos A, Papanikolaou A, Vasilagkos G, Davlouros P. Distal or Traditional Transradial Access Site for Coronary Procedures: A Single-Center, Randomized Study. JACC Cardiovasc Interv. 2022 Jan 10;15(1):22-32. doi: 10.1016/j.jcin.2021.09.037. Epub 2021 Dec 15. PMID 34922888
- [Background] Tsigkas G, Papageorgiou A, Moulias A, Apostolos A, Kalogeropoulos AP, Davlouros P. Reply: Distal Transradial Access for Primary PCI in ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2022 Apr 11;15(7):795-796. doi: 10.1016/j.jcin.2022.02.039. No abstract available. PMID 35393114
- [Background] Aminian A, Sgueglia GA, Wiemer M, Kefer J, Gasparini GL, Ruzsa Z, van Leeuwen MAH, Ungureanu C, Leibundgut G, Vandeloo B, Kedev S, Bernat I, Ratib K, Iglesias JF, Al Hage E, Posteraro GA, Pascut D, Maes F, Regazzoli D, Kakonyi K, Meijers TA, Colletti G, Krivoshei L, Lochy S, Zafirovska B, Horak D, Nolan J, Degrauwe S, Tobita K, Saito S. Distal Versus Conventional Radial Access for Coronary Angiography and Intervention: The DISCO RADIAL Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1191-1201. doi: 10.1016/j.jcin.2022.04.032. Epub 2022 May 17. PMID 35595673
- [Background] Le May M, Wells G, So D, Chong AY, Dick A, Froeschl M, Glover C, Hibbert B, Marquis JF, Blondeau M, Osborne C, MacDougall A, Kass M, Paddock V, Quraishi A, Labinaz M. Safety and Efficacy of Femoral Access vs Radial Access in ST-Segment Elevation Myocardial Infarction: The SAFARI-STEMI Randomized Clinical Trial. JAMA Cardiol. 2020 Feb 1;5(2):126-134. doi: 10.1001/jamacardio.2019.4852. PMID 31895439
- [Background] Valgimigli M, Frigoli E, Leonardi S, Vranckx P, Rothenbuhler M, Tebaldi M, Varbella F, Calabro P, Garducci S, Rubartelli P, Briguori C, Ando G, Ferrario M, Limbruno U, Garbo R, Sganzerla P, Russo F, Nazzaro M, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Ferrante G, Santarelli A, Sardella G, de Cesare N, Tosi P, van 't Hof A, Omerovic E, Brugaletta S, Windecker S, Heg D, Juni P; MATRIX Investigators. Radial versus femoral access and bivalirudin versus unfractionated heparin in invasively managed patients with acute coronary syndrome (MATRIX): final 1-year results of a multicentre, randomised controlled trial. Lancet. 2018 Sep 8;392(10150):835-848. doi: 10.1016/S0140-6736(18)31714-8. Epub 2018 Aug 25. PMID 30153988
- [Background] Xie L, Wei X, Xie Z, Jia S, Xu S, Wang K. Feasibility of Distal Radial Access for Coronary Angiography and Percutaneous Coronary Intervention: A Single Center Experience. Cardiology. 2021;146(5):531-537. doi: 10.1159/000517076. Epub 2021 Aug 6. PMID 34365454
- [Background] Kim Y, Lee JW, Lee SY, Bae JW, Lee SJ, Jeong MH, Lee SH, Ahn Y. Feasibility of primary percutaneous coronary intervention via the distal radial approach in patients with ST-elevation myocardial infarction. Korean J Intern Med. 2021 Mar;36(Suppl 1):S53-S61. doi: 10.3904/kjim.2019.420. Epub 2020 Mar 3. PMID 32122114
- [Background] Lee OH, Kim Y, Son NH, Roh JW, Im E, Cho DK, Choi D. Comparison of Distal Radial, Proximal Radial, and Femoral Access in Patients with ST-Elevation Myocardial Infarction. J Clin Med. 2021 Aug 2;10(15):3438. doi: 10.3390/jcm10153438. PMID 34362221
- [Background] Neumann F-J, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, et al. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. England; 2019;40:87-165.
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, et al. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Soci. Eur Heart J. England; 2018;39:119-77.
- [Background] Elmahdy MF, ElMaghawry M, Hassan M, Kassem HH, Said K, Elfaramawy AA. Comparison of Safety and Effectiveness Between Right Versus Left Radial Arterial Access in Primary Percutaneous Coronary Intervention for Acute ST Segment Elevation Myocardial Infarction. Heart Lung Circ. 2017 Jan;26(1):35-40. doi: 10.1016/j.hlc.2016.04.021. Epub 2016 May 25. PMID 27374862
- [Background] Hamilton GW, Sharma V, Yeoh J, Yudi MB, Raman J, Clark DJ, Farouque O. Ultrasound Guidance for Transradial Access in the Cardiac Catheterisation Laboratory: A Systematic Review of the Literature and Meta-Analysis. Heart Lung Circ. 2024 Oct;33(10):1404-1413. doi: 10.1016/j.hlc.2024.04.308. Epub 2024 Jun 12. PMID 38871531
- [Background] Soydan E, Akin M. Left Distal Radial Artery Access Site in Primary Percutaneous Coronary Intervention: Is It Safe? Balkan Med J. 2020 Aug 11;37(5):276-280. doi: 10.4274/balkanmedj.galenos.2020.2020.4.49. Epub 2020 Jun 4. PMID 32495613
- [Background] Oliveira MD, Navarro EC, Caixeta A. Distal transradial access for coronary procedures: a prospective cohort of 3,683 all-comers patients from the DISTRACTION registry. Cardiovasc Diagn Ther. 2022 Apr;12(2):208-219. doi: 10.21037/cdt-21-542. PMID 35433348
- [Background] Oliveira MDP, Navarro EC, Kiemeneij F. Distal transradial access as default approach for coronary angiography and interventions. Cardiovasc Diagn Ther. 2019 Oct;9(5):513-519. doi: 10.21037/cdt.2019.09.06. PMID 31737522
- [Background] Tsigkas G, Apostolos A, Davlouros P. Less Is More, But Not Always: Distal Transradial Access for Radial Artery Occlusion Prevention. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1202-1204. doi: 10.1016/j.jcin.2022.05.001. Epub 2022 May 17. No abstract available. PMID 35583362
- [Background] Ziakas A, Didagelos M, Hahalis G, Koutouzis M, Tsigkas G, Bompotis G, Toutouzas K, Kartalis A, Hamilos M, Kouparanis A, Sanidas E, Skalidis I, Papadopoulos T, Katranas S, Tsioufis K, Karvounis H. Characteristics of the transRADIAL approach for coronary angiography and angioplasty in GREECE: the RADIAL-GREECE registry. Hellenic J Cardiol. 2018 Jan-Feb;59(1):52-56. doi: 10.1016/j.hjc.2017.07.009. Epub 2017 Aug 12. No abstract available. PMID 28807802
- [Background] Hahalis G, Tsigkas G, Kakkos S, Panagopoulos A, Tsota I, Davlouros P, Xanthopoulou I, Koniari I, Grapsas N, Christodoulou I, Almpanis G, Leopoulou M, Kounis N, Alexopoulos D. Vascular Complications Following Transradial and Transulnar Coronary Angiography in 1600 Consecutive Patients. Angiology. 2016 May;67(5):438-43. doi: 10.1177/0003319715592095. Epub 2015 Jun 29. PMID 26124493